CLINICAL TRIAL: NCT00782106
Title: Phase 1/2 Determination of the Dose of Recominant Human Hyaluronidase (rHuPH20) Required Enabling Up to 600 mg/kg Bodyweight of IGIV, 10% to be Administered Subcutaneously in a Single Infusion Site in Subjects With Primary Immunodeficiency (PID)
Brief Title: Study to Determine the Dose of Recombinant Human Hyaluronidase Needed to Infuse a Full Dose of IGIV Subcutaneously
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160602
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tolerability of subcutaneous infusions
  Interventions: Biological: Recombinant human hyaluronidase + immune globulin intravenous
- 2 (Experimental): Tolerability of subcutaneous infusions and pharmacokinetics
  Interventions: Biological: Recombinant human hyaluronidase + immune globulin intravenous

INTERVENTIONS:
Biological: Recombinant human hyaluronidase + immune globulin intravenous — Dose (calculated) of rHuPH20 followed by subcutaneous infusion of IGIV, 10% to determine tolerability: doses of rHuPH20 and IGIV, 10% to be increased, as tolerated and as per protocol, until a full 4-week IgG dose can be administered
  Other Names: IGIV; 10% = Immune Globulin Intraveneous (Human); 10%; rHuPH20 = Recombinant Human Hyaluronidase
  Arms: 1
Biological: Recombinant human hyaluronidase + immune globulin intravenous — 1. IV infusion of IGIV, 10% to determine pharmacokinetics
  2. Intervention as in Arm 1: Dose (calculated) of rHuPH20 followed by subcutaneous infusion of IGIV, 10% to determine tolerability: doses of rHuPH20 and IGIV, 10% to be increased, as tolerated and as per protocol, until a full 4-week IgG dose can be administered
  Other Names: IGIV; 10% = Immune Globulin Intraveneous (Human); 10%; rHuPH20 = Recombinant Human Hyaluronidase
  Arms: 2

SUMMARY:
The purpose of the study is to determine the feasibility of infusing a full 4-week dose of Immune Globulin Intravenous (Human), 10% in a single subcutaneous site and the amount of recombinant human hyaluronidase needed to infuse that dose with no more than mild local adverse drug reactions.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from either the subject or the subject's legally acceptable representative
* Diagnosis of a PID disorder as defined by World Health Organization criteria1 for which the subject had been receiving a regimen of weekly or biweekly (every-other-week) subcutaneous IgG infusions or IGIV infusions every 21 to 28 days over a period of at least 8 weeks pre-study at an equivalent of a 4-week dose of 300 to 800 mg/kg bodyweight
* Adults/adolescents aged 16 years and older)
* For female subjects of child-bearing age: negative urine pregnancy test result at study entry and agreement to employ adequate birth control measures for the duration of the study

Exclusion Criteria:

* Subjects positive at enrollment for one or more of the following: HBsAg, PCR for HCV, PCR for HIV Type 1
* Subjects with levels of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal for the testing laboratory
* Subjects with neutropenia (defined as an absolute neutrophil count [ANC] <= 500/mm3).
* Subjects with serum creatinine levels greater than 1.5 times the upper limit of normal for age and gender
* Subjects with current history of malignancy
* Subjects with a history of thrombotic episodes (deep vein thrombosis, myocardial infarction, cerebrovascular accident)
* Subjects with abnormal protein loss (protein losing enteropathy, nephritic syndrome, severe lung disease)
* Subjects with anemia that in the opinion of the investigator precluded phlebotomy for laboratory studies
* Subjects who had been exposed to any blood or blood product other than an intravenous immunoglobulin (IGIV), SC immunoglobulin (SCIG), immune serum globulin (ISG) preparations, or albumin within the 6 months prior to study entry.
* Subjects with an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following IGIV, SCIG and/or ISG infusions
* Subjects with IgA deficiency and known anti IgA antibodies
* Subjects who had received antibiotic therapy for the treatment of infection within 7 days prior to enrollment
* Subjects who had participated in another clinical study involving an investigational product or device within 28 days prior to study entry
* Subjects with inability or unwillingness to meet all the requirements of this study
* If female, pregnancy or lactation at time of study entry

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-12-04 (Actual); Primary Completion 2007-11-01 (Actual); Study Completion 2007-11-01 (Actual)

PRIMARY OUTCOMES:
Ability to administer, after priming with recombinant human hyaluronidase, at least one half of a 4-week dose (minimum of 200 mg/kg) of IgG in a single infusion site, via the subcutaneous route, with no more than mild local adverse drug reactions. | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- United States (3):
  - First Allergy and Clinical Research Center, Centennial, Colorado
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Pediatrics Allergy/Immunology Association, PA, Dallas, Texas